CLINICAL TRIAL: NCT07306455
Title: Evaluatıon of the Valıdıty of a Wearable Motıon Analysıs Sensor in Assessıng Jump Heıght
Brief Title: Validity of Wearable Sensor for Jump Height
Acronym: Jump
Status: Completed | Type: Observational
Sponsor: Busra Kalkan Balak (Other)
Responsible Party: Sponsor-Investigator, Busra Kalkan Balak, Principal Investigator, PT, PhD, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Other Study IDs: AnkaraYBU-02-1155; 02-1155 (Other: Ankara Yıldırım Beyazıt University Faculty of Health Sciences Ethics Committee)
Record Dates: First submitted 2025-09-29; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers; Physical Fitness (G11.427.410.698)
Keywords: jumping; physical fitness; wearable electronic devices; validity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy female participants aged 18-35 years performed countermovement jumps. Jump height was measured simultaneously using the BTS G-sensor and the My Jump application.
  Interventions: Device: BTS G-sensor

INTERVENTIONS:
Device: BTS G-sensor — A wearable motion analysis sensor used to assess countermovement jump height.
  Other Names: my jump lab
Device: BTS G-sensor — A wearable inertial measurement unit (IMU) used to assess countermovement jump (CMJ) height.

SUMMARY:
This study aims to evaluate the concurrent validity of a wearable motion sensor (BTS G-sensor) in measuring countermovement jump (CMJ) height. Healthy female volunteers between 18 and 35 years of age will perform CMJ tests. Jump height will be measured simultaneously using the BTS G-sensor and the My Jump smartphone application, which has previously demonstrated validity and reliability. The study will assess the level of agreement between the two measurement methods.

DETAILED DESCRIPTION:
Vertical jump height is widely used as an indicator of lower limb strength and functional performance. Force platforms are the gold standard for jump height measurement but are expensive and not always practical. Wearable motion sensors and smartphone applications have been developed as low-cost and portable alternatives.

This observational study is designed to examine the concurrent validity of the BTS G-sensor, a wearable inertial measurement unit, for measuring countermovement jump (CMJ) height. Measurements obtained from the BTS G-sensor will be compared with those from the My Jump smartphone application, a validated reference tool.

Healthy female volunteers aged 18-35 years will perform countermovement jumps after a standardized warm-up. Each participant's jump height will be simultaneously recorded by both methods. Data will be analyzed using correlation and agreement analyses to determine the level of consistency between the two methods.

This is an observational validation study. Both the BTS G-sensor and the My Jump application were used simultaneously for measurement purposes only. No interventional procedure or assignment was applied to participants.

Clarification on Study Type:

This is an observational validation study. Both the BTS G-sensor and the My Jump smartphone application were used simultaneously for measurement purposes only. No participant assignment or interventional procedure was applied.

ELIGIBILITY:
* Inclusion Criteria:Female volunteers aged 18-35 years
* No history of orthopedic injury in the past 6 months
* No neurological disorders
* Not taking medications affecting balance
* Exclusion Criteria: Body Mass Index (BMI) > 25
* History of orthopedic surgery
* Impaired lower extremity joint range of motion
* Inability to complete the test protocol
* Measurement errors or missing data

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy female volunteers between the ages of 18 and 35 years were recruited from Ankara Yildirim Beyazıt University. Participants had no recent orthopedic injuries, no neurological conditions, and were not using medications that could affect balance.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Jump Height Measured with BTS G-sensor Compared to My Jump Application | single testing session, Day 1
  Countermovement jump (CMJ) height measured simultaneously with the BTS G-sensor and the My Jump smartphone application. Agreement between the two methods will be analyzed using correlation and Bland-Altman plots.
Jump Height measured with BTS G-sensor compared to My Jump application | single testing session, Day 1
  The countermovement jump (CMJ) height will be measured simultaneously using the BTS G-sensor and the My Jump smartphone application. Correlation and agreement between the two methods will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuksek İhtisas University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet determined whether individual participant data (IPD) will be shared. Decisions will depend on future institutional policies and publication requirements.

REFERENCES:
- See also: Ankara Yildirim Beyazıt University Faculty of Health Sciences — https://aybu.edu.tr/saglikbilimleri